CLINICAL TRIAL: NCT04638504
Title: Comparison of Brachial Artery Dilatation, Uterine Artery Doppler, Umbilical Artery Doppler and 1st-trimester Visceral Adipose Tissue Measurement in Obese and Normal Pregnant Women
Status: Completed | Type: Observational
Sponsor: Diyarbakir Women's and Children's Diseases Hospital (Other)
Responsible Party: Principal Investigator, Şerif AKSİN, Doctor of medicine, Diyarbakir Women's and Children's Diseases Hospital
Other Study IDs: DiyarbakirWCDH 3
Record Dates: First submitted 2020-10-18; First posted 2020-11-20 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2021-02

CONDITIONS: Obese; Vascular Diseases; Pregnancy Related; Visceral Obesity
MeSH Terms: conditions — Obesity; Vascular Diseases; Obesity, Abdominal | interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- 11-14 weeks of normal pregnancy.: 11-14. Measurement of brachial artery flow dilatation in the arm during pregnancy weeks, Visceral adipose tissue measurement (armellini method), and maternal uterine artery dopes will be examined ultrasonographically.
  Interventions: Other: ultrasonography
- 11-14 week obese pregnant: 11-14. Measurement of brachial artery flow dilatation in the arm during pregnancy weeks, Visceral adipose tissue measurement (armellini method), and maternal uterine artery dopes will be examined ultrasonographically.
  Interventions: Other: ultrasonography
- 24-28 week normal pregnant: 24-28. Measurement of brachial artery flow dilatation in the arm during pregnancy weeks, fetal umbilical artery, and maternal uterine artery dopes will be examined ultrasonographically.
  Interventions: Other: ultrasonography
- 24w-28w obese normal pregnant: 24w-28w. Measurement of brachial artery flow dilatation in the arm during pregnancy weeks, fetal umbilical artery and maternal uterine artery dopes will be examined ultrasonographically
  Interventions: Other: ultrasonography
- 37w -40w normal pregant: 37w-40 w. Measurement of brachial artery flow dilatation in the arm during pregnancy weeks, fetal umbilical artery and maternal uterine artery dopes will be examined ultrasonographically
  Interventions: Other: ultrasonography
- 37-40 w obese normal pregnant: 37w-40 w. Measurement of brachial artery flow dilatation in the arm during pregnancy weeks, fetal umbilical artery and maternal uterine artery dopes will be examined ultrasonographically
  Interventions: Other: ultrasonography

INTERVENTIONS:
Other: ultrasonography — vascular and adipose tissue measurement by ultrasonography

SUMMARY:
Brachial artery flow-mediated in obese and normal-weight pregnant women dilation of uterine artery doppler and umbilical artery doppler results comparison of

DETAILED DESCRIPTION:
The systemic inflammatory effect caused by obesity and vascular disorder It has been reported that it creates studies. Healthy Vascular Endothelial structure increases vascular tone by regulating nitric oxide (NO) release. Reduced nitric oxide production, reducing flexibility It has a facilitating effect on hypertensive diseases and other obstetric diseases.

Endothelial function, which is a non-invasive, easily applicable, and reproducible method It can be detected by endothelium-dependent vasodilation. A good indicator of endothelial function in studies in which the brachial artery flow-mediated dilation (FMD) shown. Brachial artery blood pressure cuff at forearm level in normal healthy people with compression for 3-5 minutes 50 mmHg above systolic pressure, 60-120 seconds after loosening the cuff When measured later, individuals with healthy endovascular function and the brachial artery are also reactive hyperemia, and a 10% dilatation is expected. Many obstetric effects such as obesity preeclampsia, preterm labor, gestational diabetes, preterm labor Although it was found to be related to pathology, the relationship between them could not be determined exactly.

Our study aimed to increase brachial artery dilatation in obese and normal pregnant women.

By comparing, determine the level of nitric oxide and endovascular function. Also uterine Vascular structures of obesity by comparing vascular structures with artery and umbilical uterine dops examine the effect on

Pregnant women between the ages of 18-40 who apply to the Diseases and Obstetrics outpatient clinic will be taken. 24-28. Brachial artery dilatation, uterine, and umbilical artery doppler between 11-14, 37-40w weeks between gestational weeks, and visceral adipose tissue measurement at first trimester will be examined.

ELIGIBILITY:
Inclusion Criteria:

* obese and normal pregnant
* 11-14 weeks
* 24-28 weeks
* 37-40 weeks

Exclusion Criteria:

* smoking
* chronic vascular disease
* Diabetes mellitus
* Over 40 years old

Ages: 18 Years to 40 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — pregnant
Study Population: 240
Sampling Method: Non-Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2020-11-19 (Actual); Primary Completion 2021-02-27 (Actual); Study Completion 2021-02-27 (Actual)

PRIMARY OUTCOMES:
To define the relationship between obesity and endovascular dysfunction by brachial artery dilatation method. | 3 month
  To examine the possible effects of obesity on the endovascular system with the brachial artery dilation method.
Measurement of uterine artery doppler in obese and normal pregnant women | 3 month
  To determine whether obesity has an effect on uterine artery resistance.
Measurement of obese and normal pregnant umbilical artery doppler | 3 month
  trying to understand whether obesity has fetal effects by examining umbilical artery doppler in obese pregnants and normal pregnants,
First trimester visceral adipose tissue and brachial artery measurement | 3 month
  By measuring the amount of visceral tissue in the first trimester obese and normal pregnant women with Armellini method; Investigation of its effects on endovascular dysfunction through brachial artery dilatation

CONTACTS AND LOCATIONS:
Overall Officials: Şeyhmus Tunç, MD, Study Director — Diyarbakır Gynecology Maternity and Pediatrics Hospital
Locations (1):
- Diyarbakır Women's and Children's Hospital, Diyarbakır, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adali E, Kurdoglu M, Adali F, Cim N, Yildizhan R, Kolusari A. The relationship between brachial artery flow-mediated dilatation, high sensitivity C-reactive protein, and uterine artery doppler velocimetry in women with pre-eclampsia. J Clin Ultrasound. 2011 May;39(4):191-7. doi: 10.1002/jcu.20781. Epub 2010 Dec 28. PMID 21480285
- [Background] Takase B, Goto T, Hamabe A, Uehata A, Kuroda K, Satomura K, Ohsuzu F, Kurita A. Flow-mediated dilation in brachial artery in the second half of pregnancy and prediction of pre-eclampsia. J Hum Hypertens. 2003 Oct;17(10):697-704. doi: 10.1038/sj.jhh.1001599. PMID 14504628
- [Background] Sierra-Laguado J, Garcia RG, Lopez-Jaramillo P. Flow-mediated dilatation of the brachial artery in pregnancy. Int J Gynaecol Obstet. 2006 Apr;93(1):60-1. doi: 10.1016/j.ijgo.2006.01.015. Epub 2006 Mar 9. No abstract available. PMID 16527277
- [Background] Oliveira OP, Araujo Junior E, Lima JW, Salustiano EM, Ruano R, Martins WP, Costa Fda S. Flow-mediated dilation of brachial artery and endothelial dysfunction in pregnant women with preeclampsia: a case control study. Minerva Ginecol. 2015 Aug;67(4):307-13. Epub 2014 Dec 5. PMID 25476264
- [Background] Parikh NI, Keyes MJ, Larson MG, Pou KM, Hamburg NM, Vita JA, O'Donnell CJ, Vasan RS, Mitchell GF, Hoffmann U, Fox CS, Benjamin EJ. Visceral and subcutaneous adiposity and brachial artery vasodilator function. Obesity (Silver Spring). 2009 Nov;17(11):2054-9. doi: 10.1038/oby.2009.60. Epub 2009 Mar 12. PMID 19282819